CLINICAL TRIAL: NCT00193934
Title: Prospective Study to Determine the Relationships Between Survival and FIGO Stage, Tumour Volume and Corpus Invasion in Cervical Cancer
Brief Title: Magnetic Resonance Imaging (MRI) Staging of Cervix Cancer
Status: Completed | Type: Observational
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Principal Investigator, TROG Administrator, Rebecca Montgomery, Trans Tasman Radiation Oncology Group
Other Study IDs: TROG 04.02
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Cancer of the Uterine Cervix
Keywords: Women's Health; Multidisciplinary, multicentre prospective study; Cancer:mechanisms of growth, invasion, metastases; Figo Stages cervical cancer; Advances in diagnosis using radiological methods; Quantitative Magnetic Resonance Imaging; Patient Management Strategies; Selecting patients for therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Cervical Cancer Patients

SUMMARY:
The researchers propose that it may be corpus invasion, rather than tumour volume per se, which is one of the important determinants of ultimate outcome in cervix cancer. The aim of the proposed prospective, multicentre study, is to confirm the results of our retrospective studies, specifically that corpus invasion or tumour volume or both contribute important prognostic information over and above that provided by the currently used International Federation of Gynecology and Obstetrics (FIGO) staging system. A successful outcome would have important implications for the staging, and management as well as the biologic understanding of the behaviour of cervical cancer.

DETAILED DESCRIPTION:
This will be a prospective, multicentre, prognostic factor, follow-up study. The study is designed to be as simple as possible: newly diagnosed cervical cancer patients will have key prognostic variables collected at baseline. The treatment received will be documented at the end of treatment and patients will then be followed for first relapse and survival.

Registration of a patient on this study can be undertaken after EUA, biopsy confirmed diagnosis, anatomic staging diagram and MRI have been done and before any treatment has commenced.

Treatment must be curative in intent (termed radical therapy) but otherwise can be at the discretion of the investigator. Radical hysterectomy alone, hysterectomy followed by adjuvant radiotherapy, radical chemo-radiotherapy or radical radiotherapy will be allowed. Details of the planned and given treatment regimen will be recorded.

All patients will have the following trial data documented at the time of registration:

* Age
* ECOG performance status
* smoking status
* date of histological diagnosis
* histologic type and features
* presenting haemoglobin
* standard FIGO staging
* maximum clinical tumour diameter measured at EUA
* detailed staging diagram drawn at EUA
* nodal status (by surgical pathology or CT or MRI or both and PET if available)
* date of MRI
* MRI tumour diameters
* presence or absence of corpus invasion on MRI
* planned treatment details

All patients will be assessed pre-treatment, immediately following treatment and will be followed up for local control and survival at yearly intervals from the date of registration.

It is intended to collect follow up information on all patients until one year after the final patient is registered on study.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed, biopsy proven carcinoma of the uterine cervix.
2. Squamous cell, adenocarcinoma, adenosquamous or large cell carcinoma histology.
3. FIGO Stage Ib -IVa.
4. Maximum clinical tumour diameter recorded.
5. MRI done within 30 days prior to registration.
6. Intention to treat radically
7. Treatment not yet started.
8. Written informed consent.
9. Available for follow-up.

Exclusion Criteria:

1. Lymphoma, small cell carcinoma and melanoma histology.
2. Previous hysterectomy
3. Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed cervical cancer patients, Female
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2006-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05-15 (Actual)

PRIMARY OUTCOMES:
Assess the prognostic significance, with respect to overall survival, of the factors, FIGO stage. Overall survival is defined as the date of registration to date of death from any cause. | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Adams, Study Chair — Oceania Oncology
Locations (16):
- Washington University School of Medicine, St Louis, Missouri, United States
- Australia (9):
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Royal Brisbane Hospital, Herston, Queensland
  - North Queensland Oncology Service, Townsville, Queensland
  - Premion - Tugun, Tugun, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- India (2):
  - Tata Memorial Hospital, Mumbai
  - Meenakshi Mission Hospital, Tamil Nadu
- New Zealand (3):
  - Auckland Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Narayan K, McKenzie A, Fisher R, Susil B, Jobling T, Bernshaw D. Estimation of tumor volume in cervical cancer by magnetic resonance imaging. Am J Clin Oncol. 2003 Oct;26(5):e163-8. doi: 10.1097/01.coc.0000091358.78047.b5. PMID 14528092
- [Background] Narayan K, McKenzie AF, Hicks RJ, Fisher R, Bernshaw D, Bau S. Relation between FIGO stage, primary tumor volume, and presence of lymph node metastases in cervical cancer patients referred for radiotherapy. Int J Gynecol Cancer. 2003 Sep-Oct;13(5):657-63. doi: 10.1046/j.1525-1438.2003.13026.x. PMID 14675351
- [Background] Narayan K. Arguments for a magnetic resonance imaging-assisted FIGO staging system for cervical cancer. Int J Gynecol Cancer. 2005 Jul-Aug;15(4):573-82. doi: 10.1111/j.1525-1438.2005.00128.x. PMID 16014109
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au